CLINICAL TRIAL: NCT02528825
Title: Effect-site Concentration of Remifentanil for Smooth Removal of the Double-lumen Endotracheal Tube
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Yoo, clinical assistant professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: AJIRB-MED-CT4-14-295
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Remifentanil Concentration for Smooth Emergence

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- smooth emergence (Experimental): ASA I-II, aged 19-65 years undergoing general anesthesia with DLT for lung wedge resection were enrolled in this study.After completing the surgery, the propofol infusion was stopped, and effect-site concentration of remifentanil was titrated to predetermined concentration ( initial concentration being 1.5ng/ml for the first patient).The predetermined concentration was maintained at least 10 min throughout emergence for the effect site concentration and plasma concentration can be expected stable. The smooth emergence was defined as extubation without cough-a strong and sudden contraction of the abdomen. The predetermined concentration was decreased by 0.5 ng/ml for the next patient if the patient did not cough during emergence and similarly, if the patient coughed anytime during emergence, it was considered failed smooth emergence and predetermined concentration was increased by 0.5 ng/ml.
  Interventions: Drug: Remifentanil titration

INTERVENTIONS:
Drug: Remifentanil titration — Initial concentration being 1.5ng/ml for the first patient The smooth emergence was defined as extubation without cough-a strong and sudden contraction of the abdomen. The predetermined concentration was decreased by 0.5 ng/ml for the next patient if the patient did not cough during emergence and similarly, if the patient coughed anytime during emergence, it was considered failed smooth emergence and predetermined concentration was increased by 0.5 ng/ml.

SUMMARY:
Smooth emergence is important for patient safety and satisfaction. Coughing during emergence is associated with detrimental effects like laryngospasm, sore throat, hoarseness, negative pressure pulmonary edema and bleeding at surgical site 1. Especially sore throat and hoarseness are most common complications after extubation 2,3 and closely related to patient satisfaction 4. Using double lumen tube (DLT) increase the incidence of hoarseness and airway injury than using single lumen tube for it has large size5,6. Various technique and drugs have been proposed for reducing coughing during extubation including smooth emergence 1,7-11 and this is closely correlate with reducing sore throat and hoarseness 12. One of the proposed technique, the use of short acting opioids are prefered13-15 because it can be maintained during emergence with less respiratory depression. Remifentanil is a potent short acting opioid and several studies choose remifentanil combined with other anesthetic agents 1,15,16. There is a study about the EC50 and EC95 of remifentanil in effect site Target controlled infusion(TCI) for preventing cough during emergence after thyroidectomy with propofol-remifentanil anesthesia 15 but no study about the proper dose of remifentanil for smooth DLT extubation.

The purpose of this study was to evaluate the EC50 and EC95 of remifentanil in effect-site TCI for preventing cough during extubation of DLT in total TIVA with propofol and remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II,
* Undergoing general anesthesia with DLT for lung wedge resection

Exclusion Criteria:

* Anticipated difficult airway
* Surgical duration of > 120 min,
* Patient with gastroesophageal reflux or asthma, chronic obstructive disease and upper respiratory infection were excluded from the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Smooth emergence success or fail | from the time of remifentanil equivalent state( postop 5 minute) to extubation
  smooth emergence is success

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Yoo, md, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Jiyoung Yoo, Suweon, Kyunggido, South Korea